CLINICAL TRIAL: NCT07392840
Title: Postoperative Delayed Neurocognitive Recovery in Elderly Patients Undergoing Spinal Anesthesia: Assessment of Its Prevalence and Correlation With Preoperative Sleep Disorders and Melanin Concentrating Hormone.
Brief Title: Postoperative Cognitive Dysfunction in Elderly and it's Relation With Sleep Disorders and Melanin Concentrating Hormone
Status: Not yet recruiting | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohamed Yasein Mohamed Moawad, Principal investigator, assistant lecturer anesthesiologist, Minia University
Other Study IDs: Postop. cognitive dysfunction
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: 25 patients with preoperative sleep disorders
- Group B: 25 patients without preoperative sleep disorders

SUMMARY:
The aim of this study is to explore the relationship between preoperative sleep disorders, melanin-concentrating hormone (MCH), and delayed neurocognitive recovery early after surgery in older adult patients undergoing spinal anesthesia.

DETAILED DESCRIPTION:
Perioperative neurocognitive disorders (PNDs) have gradually become a priority during the perioperative period, including neurocognitive disorder before surgery, delirium and delayed neurocognitive recovery (DNR) within 30 days after surgery, and postoperative neurocognitive disorder up to 12 months after surgery. The incidence of DNR ranges from 9.1% to 45%, which seriously affects the perioperative brain health of older adult patients .

The increasing aging population and the reduced function and compensatory capacity of various systems in elderly patients also significantly increase the risk of cognitive dysfunction .

Sleep disorders are critical risk factors among the various risk factors for DNR after surgery. Meanwhile, aging is an independent risk factor for sleep disorders .

Therefore, it is clinically significant to conduct early cognitive risk prediction, focusing on older adult patients with preoperative sleep disorders. Studies have explored the risk factors for perioperative sleep disorders, while other studies have also explored the risk factors affecting postoperative cognitive outcomes. However, no study has explored the specific risk factors for DNR in patients with preoperative sleep disorders. Considering the relationship between sleep and postoperative cognitive function, especially in older adult patients, it is necessary to link these 2 main risk factors (preoperative sleep disorders and DNR) that impair the perioperative brain health to explore potential biomarkers .

Melanin-concentrating hormone (MCH) is a highly conserved cyclic neuropeptide with 19 amino acids in mammals and has a variety of physiological functions, including orexigenic properties, energy homeostasis, regulation of moods, sleep, wakefulness, and cognitive functions .

Melanin-concentrating hormone (MCH) can enhance synaptic plasticity in the hippocampus, which plays an important role in maintaining cognitive function In addition to regulating synaptic plasticity, MCH can also regulate cognitive functions such as learning and memory by regulating rapid eye movement (REM) sleep and acetylcholine outflow in the hippocampus .

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders ageing 65 years or above.
* ASA grade I to III.
* Undergo elective lower limb surgery under spinal anesthesia
* Agree to collect one's own CSF and blood samples

Exclusion Criteria:

* Past history of depression,anxiety,delirium and schizophrenia .
* Past history of drug dependence.
* Past history of dementia,including Alzheimer disease(AD).
* Preoperative Montreal Cognitive Assessment (MoCA) score <26.
* Inability to understand or cooperate with the evaluation scale or questionnaire.
* Refuse collecting one's own CSF and blood samples.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A total of (50) patients candidate for elective lower limb surgery aged from 65 years of both sexes will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the impact of preoperative sleep problems as indicators of delayed neurocognitive recovery (DNR) in elderly adults following spinal anesthesia. | Baseline, one week, three months
  By comparison between the two groups

SECONDARY OUTCOMES:
to investigate the predictive power of CSF and plasma MCH levels for delayed neurocognitive recovery (DNR) in older adults after spinal anesthesia | Baseline one day before operation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mostafa Ali, MD, Principal Investigator — El-minya University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner S, Ahrens E, Wachtendorf LJ, et al. Association of obstructive sleep apnea with postoperative delirium in procedures of moderate-to-high complexity: a hospital-registry study. Anesth Analg. 2023.
- [Background] Travica N, Lotfaliany M, Marriott A, et al. Peri-operative risk factors associated with post-operative cognitive dysfunction (POCD): an umbrella review of meta-analyses of observational studies. J Clin Med. 2023;12:1610.
- [Background] POIRIER, Gabriel, et al. Deterioration, compensation and motor control processes in healthy aging, mild cognitive impairment and Alzheimer's disease. Geriatrics, 2021, 6.1: 33
- [Background] Monti JM, Torterolo P, Lagos P. Melanin-concentrating hormone control of sleep-wake behavior. Sleep Med Rev.2013;17:293-298. Nasreddine ZS, Phillips NA, Bedirian V, et al. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005;53:695-699.
- [Background] Li Yun,Zhang Xizhe, et al . Research progress on the role of melanin-concentrating hormone system in sleep deprivation -induced impairment of learning and memory function [ J ] . International Journal of Anesthesiology and Resuscitation , 2022 , 43 ( 10 ): 1117-1120 .
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res.1989;28:193-213.
- [Background] Butris N, Tang E, Pivetta B, et al. The prevalence and risk factors of sleep disturbances in surgical patients:a systematic review and meta-analysis. Sleep Med Rev.2023;69:101786.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, et al. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005;53:695-699.
- [Background] Monti JM, Torterolo P, Lagos P. Melanin-concentrating hormone control of sleep-wake behavior. Sleep Med Rev.2013;17:293-298.